CLINICAL TRIAL: NCT07137039
Title: A Single-arm, Prospective, Single-center Clinical Study on Neoadjuvant Treatment of Locally Advanced Hypopharyngeal Cancer With Adebrelimab Combined With TP Chemotherapy Regimen
Brief Title: Neoadjuvant Treatment of Locally Advanced Hypopharyngeal Cancer With Adebrelimab Combined With TP Chemotherapy Regimen
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, San-Gang Wu, Clinical Professor, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMHNC-001
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Hypopharyngeal Cancer
Keywords: hypopharyngeal cancer; neoadjuvant treatment; adebrelimab; chemotherapy
MeSH Terms: conditions — Hypopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Adebrelimab combined with albumin, paclitaxel and cisplatin
  Interventions: Drug: Adebrelimab+Albumin paclitaxel +Cisplatin

INTERVENTIONS:
Drug: Adebrelimab+Albumin paclitaxel +Cisplatin — 1. Adebrelimab：1200mg, ivgtt, D1, Q3W;
  2. Albumin paclitaxel :260mg/m2, ivgtt, D1, Q3W;
  3. Cisplatin :60mg/m2, ivgtt, D1, Q3W.

SUMMARY:
To evaluate the efficacy and safety of adebrelimab combined with TP chemotherapy regimen as neoadjuvant therapy for locally advanced hypopharyngeal cancer

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 70 years old, gender not limited;
* 2.ECOG PS score: 0-1 point;
* 3. Patients who are capable of surgical resection and willing to undergo it;
* 4. Hypopharyngeal cancer diagnosed by histology/cytology and imaging, with a clinical stage of T1-2, N1-3 or T3-4, any N;
* 5. At least one measurable lesion (in accordance with RECIST 1.1 standard);
* 6. The expected survival period is at least 12 weeks;
* 7. Other major organs (liver, kidneys, blood system, etc.) function well: Hemoglobin ≥90g/L (no blood transfusion, no use of hematopoietic factors and no drug correction within 2 weeks before the first administration); Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count ≥100×10^9/L; Total bilirubin ≤1.5 times the upper limit of the normal value; Alanine aminotransferase, aspartate aminotransferase and alkaline phosphatase ≤2.5 times the upper limit of the normal value; Serum creatinine ≤1.5 times the upper limit of the normal value, and endogenous creatinine clearance rate ≥60ml/min; For patients who have not received anticoagulant therapy, the international normalized ratio of prothrombin time (INR) is ≤1.5, and the activated partial thromboplastin time (APTT) is ≤1.5 times the upper limit of the normal value.
* 8. Female subjects with fertility must undergo a pregnancy test (serum or urine) within 72 hours before the start of the study medication, and the result must be negative. They must also be willing to use a medically approved efficient contraceptive measure (such as an intrauterine device, contraceptive pill or condom) during the study period and within 90 days after the last administration of the study drug. For male subjects whose partners are women of childbearing age, they must agree to use effective contraception or have undergone surgical sterilization during the study period and within 90 days after the last administration of the study.
* 9. There is no history of allergy to related drug components.
* 10. The subjects voluntarily joined this clinical study and signed the informed consent form.

Exclusion Criteria:

* 1. Have received any anti-tumor treatment in the past, including radiotherapy, chemotherapy, targeted therapy, immunotherapy and traditional Chinese medicine anti-tumor treatment (except for the treatment of malignant tumors that have been completely cured in the past and have no recurrence or metastasis for ≥5 years);
* 2. Have undergone surgical operations targeting the primary tumor or lymph nodes in the past;
* 3. Patients who have suffered from any malignant tumors in the past five years (except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix);
* 4. Patients with distant metastases;
* 5. Suffering from any active autoimmune disease or a history of autoimmune diseases (such as uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy), tuberculosis) Patients with childhood asthma that has been completely relieved and do not require any intervention or systemic treatment in adulthood (such as vitiligo, psoriasis or alopecia) can be included. However, patients who need medical intervention with bronchodilators cannot be included.
* 6. Subjects who have received systemic treatment with corticosteroids (prednisone or other equivalent hormones >10 mg/ day) or other immunosuppressants within 2 weeks prior to the first administration. In the absence of active autoimmune diseases, inhalation or topical use of corticosteroids, as well as adrenal hormone replacement therapy with a dose of ≤10 mg/ day at the therapeutic dose of prednisone, is permitted.
* 7. Those who have experienced hyperactive or venous thrombosis events within 6 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
* 8. Within 3 months prior to enrollment, significant clinically significant bleeding symptoms or a clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc., have occurred, or are currently receiving thrombolytic or anticoagulant therapy;
* 9. Those with hypertension who have not achieved good control through antihypertensive drug treatment (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); Or grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥450ms in men and ≥470ms in women); According to the NYHA standard, patients with grade Ⅲ to Ⅳ cardiac failure, or those whose left ventricular ejection fraction (LVEF) is less than 50% as indicated by echocardiography;
* 10. Urine routine test indicates urine protein ≥(++), or 24-hour urine protein content ≥1g, or severe liver and kidney dysfunction;
* 11. Allergic to the test drug;
* 12. Known human immunodeficiency virus (HIV) infection;
* 13. Pregnant or lactating women; Subjects with fertility who are unwilling or unable to take effective contraceptive measures;
* 14. Those who suffer from neurological or mental disorders and are unable to cooperate;
* 15. Other circumstances that the researchers consider unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-08-20 (Estimated); Study Completion 2028-08-20 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | Six months
  Pathological examination of the resected tissue samples did not reveal any residual tumor cells.

SECONDARY OUTCOMES:
Major pathological response (MPR) | six months
  Major pathological response (MPR) is defined as the presence of active tumor tissue in surgical specimens ≤10% at the time of tumor resection.
Surgical R0 resection rate | Six months
  The proportion of the resection margin without residual cancer cells
Laryngeal function retention rate | six months
  It refers to the proportion of subjects whose laryngeal functions (including vocalization, breathing and swallowing functions) are successfully preserved during the treatment process through methods such as surgery, radiotherapy, chemotherapy or comprehensive treatment.
The intensity of the surgery has decreased | six months
  The researchers determined whether the surgical intensity had decreased based on the subjects' conditions.
Objective response rate (ORR) | one year
  It refers to the proportion of all subjects whose best overall response (BOR) was rated as complete response (CR) or partial response (PR) according to the RECIST 1.1 standard.
Disease Control rate (DCR) | One year
  It refers to the proportion of all subjects whose overall response rate (BOR) was rated as complete response (CR), partial response (PR), and stable disease (SD) according to the RECIST 1.1 standard.
Recurrence-free survival time (RFS) | Two years
  It refers to the period from the date of successful surgery to recurrence or death.
Overall survival (OS) | Two years
  Defined as the period from the date of the first administration to the death of the subject for various reasons.
Adverse event(AE) | Two years
  The incidence and severity of adverse events (AE) evaluated according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No